CLINICAL TRIAL: NCT05815069
Title: Clinical Study of Chemokine Receptor 4 (CXCR4)-Mediated Precision Targeting of 18F for the Diagnosis of Aldosteronism in Primary Aldosteronism
Brief Title: [18F]AlF-NOTA-pentixather PET/CT in Patients With Suspected Primary Hyperaldosteronism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Hao Wang, Associate senior physician, Sichuan Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SCPHNM2
Record Dates: First submitted 2023-03-22; First posted 2023-04-18 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Aldosterone-Producing Adenoma
MeSH Terms: conditions — Adrenocortical Adenoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [18F]AlF-NOTA-pentixather (Experimental): No special preparation such as fasting and fasting is required before the examination. The radiotracer 18F-AlF-NOTA-pentiaxther PET/CT (dose 4.81 MBq/Kg body weight) was injected intravenously according to the patient's body weight, and the drug was synthesized by the Department of Nuclear Medicine of Sichuan Provincial People's Hospital immediately before the examination. Before the examination, patients were instructed to urinate as many times as possible to reduce the possible influence of the residual radiotracer in the renal pelvis and calyces on the image quality. The whole-body PET/CT examination from the top of the skull to the root of the thigh was performed using a PET/CT examination instrument (Siemens Biograph mCT Flow) 50-60 minutes after the injection of radiopharmaceuticals. Flow Motion flow scanning technology with a matrix of 128x128 and a layer thickness of 3 mm was used. all PET images were reconstructed iteratively.
  Interventions: Diagnostic Test: [18F]AlF-NOTA-pentixather PET/CT

INTERVENTIONS:
Diagnostic Test: [18F]AlF-NOTA-pentixather PET/CT — The radiotracer 18F-AlF-NOTA-pentixather PET/CT (dose 4.81 MBq/Kg body weight) was injected intravenously according to the patient's body weight. The whole-body PET/CT examination from the top of the skull to the root of the thigh was performed using a PET/CT examination instrument (Siemens Biograph mCT Flow) 50-60 minutes after the injection of radiopharmaceuticals. Flow Motion flow scanning technology with a matrix of 128x128 and a layer thickness of 3 mm was used. all PET images were iteratively reconstructed. Patients who have undergone surgery routinely undergo pathological examination.
  Other Names: pathological examination

SUMMARY:
The study was proposed to include 20 patients with clinical suspicion of primary aldosteronism for [18F]AlF-NOTA-pentixather PET/CT imaging and to analyze the specificity and sensitivity of [18F]AlF-NOTA-pentixather PET/CT for the diagnosis of APA by comparison with the final pathological findings.

ELIGIBILITY:
Inclusion Criteria:

* Persistent hypertension or refractory hypertension (blood pressure >140/90 mmHg with a combination of three antihypertensive drugs, including diuretics) with hypokalemia of blood pressure >160/100 mmHg.
* Uncontrollable hypokalemia with or without hypertension. Persistent hypertension or refractory hypertension with blood pressure >160/100 mmHg and aldosterone-renin ratio (ARR) ≥30 (ng/dl)/(ng/ml/h).
* Positive captopril test (≤30% decrease in plasma aldosterone level after captopril administration) is a sufficient but not mandatory condition.
* Patients with CT showing unilateral or bilateral adrenal nodules with well-defined borders but normal serum potassium and ARR <30 (ng/dl)/(ng/ml/h) were also included in the study.

Exclusion Criteria:

* Female patients who are pregnant (or intend to become pregnant within six months), breastfeeding, or unwilling to use contraception.
* Abnormal cardiopulmonary function or mental status, unable to tolerate prone for 20 minutes.
* Refusal to sign an informed consent form or inability or unwillingness to comply with the investigator-approved study protocol.
* Other conditions deemed by the investigator to be inappropriate for participation in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-07 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Maximum standardized uptake value(SUVmax) | Within a week of completion of imaging
  Maximum standardized uptake value of suspicious adrenal lesion on [18F]AlF-NOTA-pentixather PET/CT
target background ratio(TBR) | Within a week of completion of imaging
  The ratio of SUVmax of adrenal lesions to SUVmean of the liver background and the ratio of SUVmax of adrenal lesions to SUVmean of the contralateral adrenal gland were analyzed in the study as the target background ratio(TBR).

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhang, Ph.D, Study Chair — Sichuan Academy of Medical Sciences
Locations (1):
- Sichuan Academy of Medical Sciences.Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ding J, Zhang Y, Wen J, Zhang H, Wang H, Luo Y, Pan Q, Zhu W, Wang X, Yao S, Kreissl MC, Hacker M, Tong A, Huo L, Li X. Imaging CXCR4 expression in patients with suspected primary hyperaldosteronism. Eur J Nucl Med Mol Imaging. 2020 Oct;47(11):2656-2665. doi: 10.1007/s00259-020-04722-0. Epub 2020 Mar 23. PMID 32206838
- [Result] Poschenrieder A, Osl T, Schottelius M, Hoffmann F, Wirtz M, Schwaiger M, Wester HJ. First 18F-Labeled Pentixafor-Based Imaging Agent for PET Imaging of CXCR4 Expression In Vivo. Tomography. 2016 Jun;2(2):85-93. doi: 10.18383/j.tom.2016.00130. PMID 30042959
- [Result] Heinze B, Fuss CT, Mulatero P, Beuschlein F, Reincke M, Mustafa M, Schirbel A, Deutschbein T, Williams TA, Rhayem Y, Quinkler M, Rayes N, Monticone S, Wild V, Gomez-Sanchez CE, Reis AC, Petersenn S, Wester HJ, Kropf S, Fassnacht M, Lang K, Herrmann K, Buck AK, Bluemel C, Hahner S. Targeting CXCR4 (CXC Chemokine Receptor Type 4) for Molecular Imaging of Aldosterone-Producing Adenoma. Hypertension. 2018 Feb;71(2):317-325. doi: 10.1161/HYPERTENSIONAHA.117.09975. Epub 2017 Dec 26. PMID 29279316